CLINICAL TRIAL: NCT02429154
Title: Assessment of Cerebral Vasoreactivity Using Near-infrared Spectroscopy (NIRS) in Infants
Brief Title: Assessment of Cerebral Vasoreactivity Using Near-infrared Spectroscopy (NIRS) in Infants (VARO)
Acronym: VARO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walid HABRE (Other)
Responsible Party: Sponsor-Investigator, Walid HABRE, Associated Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-204
Record Dates: First submitted 2015-03-11; First posted 2015-04-29 (Estimated); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Hypercapnia
Keywords: spectroscopy, near-infrared; Infant; Anesthesia, general
MeSH Terms: conditions — Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normocapnia (Active Comparator): The Child will be ventilated in order to achieve an end-tidal carbon dioxide (ETCO2) of 5.5 kiloPascal (kPa). Measurements will be performed after steady state condition. Then the ventilation will be reduced to allow ETCO2 to reach 6.5 kPa before repeating the measurements. Finally, the child will be again ventilated to obtain a normocapnia condition.
  Interventions: Other: Normocapnia
- Mild Hypercapnia (Other): The Child will be ventilated in order to achieve a ETCO2 of 6.5 kPa. Measurements will be performed after steady state condition. Then the ventilation will be increased to allow ETCO2 to reach 5.5 kPa before repeating the measurements. Finally, the child will be again ventilated to obtain a mild hypercapnic condition
  Interventions: Other: Mild Hypercapnia

INTERVENTIONS:
Other: Normocapnia — Normoventilation in order to have an end-tidal carbon dioxide (ETCO2) of 5.5 kiloPascal (kPa)
  Arms: Normocapnia
Other: Mild Hypercapnia — Decrease in minute ventilation in order to increase ETCO2 to 6.5 kPa
  Arms: Mild Hypercapnia

SUMMARY:
The purpose of this study is to show that a permissive hypercapnia during mechanical ventilation in children under general anaesthesia will improve cerebral perfusion.

DETAILED DESCRIPTION:
Mechanical ventilation interferes with cerebral perfusion via the changes in intrathoracic pressure and/or as a consequence of hypocapnia. This latter occurs frequently following traditional ventilation strategies with relatively high tidal volume and respiratory rate. New trends in anesthesia intend to promote protective lung ventilation by keeping a normocapnic or even mildly hypercapnic state. However, cerebral vascular vasotonicity is carbon dioxide (CO2)-dependent with hypocapnia potentially leading to vasoconstriction and subsequent decrease in cerebral blood flow. Changes in cerebral vasoreactivity can be assessed by the near infrared spectroscopy (NIRS) device. This monitoring evaluates the changes in various parameters (deoxygenated hemoglobin, oxygenated hemoglobin, the tissue oxygenation index (TOI) and the tissue hemoglobin index (THI)) that act as surrogate for cerebral vasoconstriction.

We, therefore designed this prospective observational comparative effectiveness study in order to characterize the potential beneficial effect of permissive hypercapnia on cerebral perfusion in infants.

ELIGIBILITY:
Inclusion Criteria:

* term neonates during their infancy
* for elective surgery requiring general anesthesia and endotracheal intubation

Exclusion Criteria:

* all infants with cardiac anomalies, chronic pulmonary disease (bronchopulmonary dysplasia, cystic fibrosis, asthma), pulmonary hypertension or cranial hypertension will be excluded
* all infants where no access to the forehead is possible as a consequence of the operating field

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2017-09 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Assessment of the changes in TOI and THI as measured by NIRS under normocapnia and permissive hypercapnia | At steady state (2-3 minutes) after achieving each level of ETCO2 and every 2 minutes up to 6 minutes for each level

SECONDARY OUTCOMES:
Blood gas analysis | 5 or 20 minutes after reaching the steady state with ETCO2
  Assessment changes in oxygen partial pressure (PaO2), carbon dioxide partial pressure (PaCO2) and potential of hydrogen (pH) under one level of ETCO2
Blood Pressure | At steady state (2-3 minutes) after achieving each level of ETCO2 and every 2 minutes up to 6 minutes for each level
  Non invasive monitoring of blood pressure
Heart rate | At steady state (2-3 minutes) after achieving each level of ETCO2 and every 2 minutes up to 6 minutes for each level
  Non invasive recording of heart rate
Body temperature | At steady state (2-3 minutes) after achieving each level of ETCO2 and every 2 minutes up to 6 minutes for each level
  Naso-pharyngeal temperature probe

CONTACTS AND LOCATIONS:
Overall Officials: Walid Habre, MD, PhD, Principal Investigator — University of Geneva
Locations (1):
- Geneva Children's Hospital, Geneva, Switzerland

REFERENCES:
- [Derived] Schopfer L, Habre W, Pichon I, Fodor GH. Effect of Permissive Mild Hypercapnia on Cerebral Vasoreactivity in Infants: A Randomized Controlled Crossover Trial. Anesth Analg. 2021 Oct 1;133(4):976-983. doi: 10.1213/ANE.0000000000005325. PMID 33410612